CLINICAL TRIAL: NCT03928704
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Bimekizumab in Subjects With Active Nonradiographic Axial Spondyloarthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Subjects With Active Nonradiographic Axial Spondyloarthritis
Acronym: BE MOBILE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS0010; 2017-003064-13 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Nonradiographic Axial Spondyloarthritis
Keywords: Nonradiographic axial spondyloarthritis; Axial spondyloarthritis; Nr-axSpA; Bimekizumab
MeSH Terms: conditions — Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis | interventions — bimekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bimekizumab (Experimental): Subjects randomized to this arm will receive bimekizumab during the Double-Blind Treatment Period and the Maintenance Period.
  Interventions: Drug: Bimekizumab
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive placebo during the Double-Blind Treatment Period and receive bimekizumab during the Maintenance Period.
  Interventions: Drug: Bimekizumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-specified time-points.
  Other Names: BKZ; UCB4940
Other: Placebo — Subjects will receive placebo at pre-specified time-points during the Double-Blind Treatment Period.
  Other Names: PBO
  Arms: Placebo

SUMMARY:
The purpose of the study is to demonstrate the efficacy, safety and tolerability of bimekizumab administered subcutaneously (sc) compared to placebo in the treatment of subjects with active nonradiographic axial spondyloarthritis (nr-axSpA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age
* Patient has nonradiographic axial spondyloarthritis (nr-axSpA) with all of the following criteria:

  1. Adult-onset axial spondyloarthritis meeting Assessment of SpondyloArthritis International Society (ASAS) classification criteria
  2. Inflammatory back pain for at least 3 months
  3. Age at symptom onset of less than 45 years
  4. NO sacroiliitis (in Anterior-Posterior pelvis or sacroiliac x-ray)
* Active disease defined by Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) >=4 AND spinal pain >=4 on a 0 to 10 Numeric Rating Scale
* Objective inflammation defined by sacroiliitis on magnetic resonance imaging and/or elevated C-reactive protein
* Subjects had to have either failed to respond to 2 different nonsteroidal anti-inflammatory drugs (NSAIDs) given at the maximum tolerated dose for a total of 4 weeks or have a history of intolerance to or a contraindication to NSAID therapy
* Patients who have taken a tumor necrosis factor alpha (TNFα) inhibitor must have experienced an inadequate response or intolerance to treatment given at an approved dose for at least 12 weeks
* Patients currently taking NSAIDs, cyclooxygenase 2 (COX-2) inhibitors, analgesics, corticosteroids, methotrexate (MTX), leflunomide (LEF), sulfasalazine (SSZ), hydroxychloroquine (HCQ) AND/OR apremilast can be allowed if they fulfill specific requirements prior to study entry

Exclusion Criteria:

* Treatment with more than 1 TNFα inhibitor and/or more than 2 additional non-TNFα biological response modifiers, or any interleukin (IL)-17 biological response modifier
* Active infection or history of recent serious infections
* Viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Any live (includes attenuated) vaccination within the 8 weeks prior to entering the study or TB (Bacillus Calmette-Guerin) vaccination within 1 year prior entering the study
* Known tuberculosis (TB) infection, at high risk of acquiring TB infection, or current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma or in situ cervical cancer
* Diagnosis of inflammatory conditions other than axial spondyloarthritis (axSpA), including but not limited to psoriatic arthritis, rheumatoid arthritis, sarcoidosis, systemic lupus erythematosus, and reactive arthritis. Patients with a diagnosis of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease (IBD) are allowed as long as they have no active symptomatic disease when entering the study
* Presence of active suicidal ideation, or moderately severe major depression or severe major depression
* Female patients who are breastfeeding, pregnant, or planning to become pregnant during the study
* Subject has a history of chronic alcohol or drug abuse within 6 months prior to Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (83):
- United States (14):
  - As0010 50131, Mesa, Arizona
  - As0010 50052, Phoenix, Arizona
  - As0010 50062, Sun City, Arizona
  - As0010 50060, Upland, California
  - As0010 50059, Ormond Beach, Florida
  - As0010 50056, Sarasota, Florida
  - As0010 50015, Hagerstown, Maryland
  - As0010 50016, St Louis, Missouri
  - As0010 50055, Portland, Oregon
  - As0010 50020, Duncansville, Pennsylvania
  - As0010 50012, Memphis, Tennessee
  - As0010 50057, Dallas, Texas
  - As0010 50036, Mesquite, Texas
  - As0010 50061, Spokane, Washington
- Belgium (4):
  - As0010 40004, Brussels
  - As0010 40003, Genk
  - As0010 40001, Ghent
  - As0010 40002, Merksem
- Bulgaria (4):
  - As0010 40006, Plovdiv
  - As0010 40007, Plovdiv
  - As0010 40005, Sofia
  - As0010 40008, Sofia
- China (9):
  - As0010 20040, Beijing
  - As0010 20021, Chengdu
  - As0010 20019, Guangzhou
  - As0010 20034, Hefei
  - As0010 20024, Nanjing
  - As0010 20018, Shanghai
  - As0010 20020, Shanghai
  - As0010 20026, Shanghai
  - As0010 20025, Wenzhou
- Czechia (8):
  - As0010 40011, Brno
  - As0010 40009, Pardubice
  - As0010 40013, Prague
  - As0010 40014, Prague
  - As0010 40015, Prague
  - As0010 40016, Prague
  - As0010 40010, Uherské Hradiště
  - As0010 40012, Zlín
- France (2):
  - As0010 40018, Boulogne-Billancourt
  - As0010 40022, Limoges
- Germany (6):
  - As0010 40025, Berlin
  - As0010 40029, Hamburg
  - As0010 40024, Hanover
  - As0010 40027, Herne
  - As0010 40078, Leipzig
  - As0010 40026, Ratingen
- Hungary (4):
  - As0010 40032, Debrecen
  - As0010 40031, Szeged
  - As0010 40033, Székesfehérvár
  - As0010 40080, Szombathely
- Japan (11):
  - As0010 20030, Chūōku
  - As0010 20039, Iruma-gun
  - As0010 20036, Kawachi-Nagano
  - As0010 20045, Kita-gun
  - As0010 20065, Kitakyushu
  - As0010 20038, Nankoku-shi
  - As0010 20037, Osaka
  - As0010 20084, Saga
  - As0010 20048, Saitama
  - As0010 20031, Sapporo
  - As0010 20035, Tokyo
- Poland (8):
  - As0010 40038, Elblag
  - As0010 40042, Krakow
  - As0010 40037, Lublin
  - As0010 40044, Poznan
  - As0010 40040, Torun
  - As0010 40041, Warsaw
  - As0010 40039, Wroclaw
  - As0010 40043, Wroclaw
- Spain (5):
  - As0010 40045, A Coruña
  - As0010 40046, Córdoba
  - As0010 40047, Madrid
  - As0010 40048, Santiago de Compostela
  - As0010 40049, Seville
- Turkey (Türkiye) (4):
  - As0010 40052, Ankara
  - As0010 40053, Ankara
  - As0010 40050, Istanbul
  - As0010 40051, Izmir
- United Kingdom (4):
  - As0010 40057, Edinburgh
  - As0010 40056, Leeds
  - As0010 40054, London
  - As0010 40055, Norwich

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] van der Heijde D, Deodhar A, Baraliakos X, Brown MA, Dobashi H, Dougados M, Elewaut D, Ellis AM, Fleurinck C, Gaffney K, Gensler LS, Haroon N, Magrey M, Maksymowych WP, Marten A, Massow U, Oortgiesen M, Poddubnyy D, Rudwaleit M, Shepherd-Smith J, Tomita T, Van den Bosch F, Vaux T, Xu H. Efficacy and safety of bimekizumab in axial spondyloarthritis: results of two parallel phase 3 randomised controlled trials. Ann Rheum Dis. 2023 Apr;82(4):515-526. doi: 10.1136/ard-2022-223595. Epub 2023 Jan 17. PMID 36649967
- [Result] Navarro-Compan V, Ramiro S, Deodhar A, Mease PJ, Rudwaleit M, de la Loge C, Fleurinck C, Taieb V, Morup MF, Massow U, Kay J, Magrey M. Association of clinical response criteria and disease activity levels with axial spondyloarthritis core domains: results from two phase 3 randomised studies, BE MOBILE 1 and 2. RMD Open. 2024 Apr 10;10(2):e004040. doi: 10.1136/rmdopen-2023-004040. PMID 38599650
- [Result] Dubreuil M, Navarro-Compan V, Boonen A, Gaffney K, Gensler LS, de la Loge C, Vaux T, Fleurinck C, Massow U, Taieb V, Morup MF, Deodhar A, Rudwaleit M. Improved physical functioning, sleep, work productivity and overall health-related quality of life with bimekizumab in patients with axial spondyloarthritis: results from two phase 3 studies. RMD Open. 2024 Jun 4;10(2):e004202. doi: 10.1136/rmdopen-2024-004202. PMID 38834351
- [Result] Cella D, de la Loge C, Fofana F, Guo S, Ellis A, Fleurinck C, Massow U, Dougados M, Navarro-Compan V, Walsh JA. The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) scale in patients with axial spondyloarthritis: psychometric properties and clinically meaningful thresholds for interpretation. J Patient Rep Outcomes. 2024 Aug 12;8(1):92. doi: 10.1186/s41687-024-00769-x. PMID 39133438
- [Result] Ramiro S, Poddubnyy D, Mease PJ, Lopez-Medina C, Kim M, Massow U, Taieb V, Kragstrup TW, McGonagle D. Sustained resolution of enthesitis and peripheral arthritis over 104 weeks with bimekizumab in axial spondyloarthritis. RMD Open. 2025 Oct 22;11(4):e005969. doi: 10.1136/rmdopen-2025-005969. PMID 41125403
- [Derived] Marzo-Ortega H, Navarro-Compan V, Dubreuil M, Mease PJ, Magrey M, Rudwaleit M, D'Agostino MA, Gaffney K, Kay J, de la Loge C, Massow U, Taieb V, Vaux T, Deodhar A. Sustained improvements in spinal pain, morning stiffness, fatigue, sleep, physical function and overall health-related quality of life with bimekizumab in patients with axial spondyloarthritis: 2-year results from two phase 3 studies. RMD Open. 2025 Nov 28;11(4):e006013. doi: 10.1136/rmdopen-2025-006013. PMID 41314667
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Navarro-Compan V, Rudwaleit M, Dubreuil M, Magrey M, Marzo-Ortega H, Mease PJ, Walsh JA, Dougados M, de la Loge C, Fleurinck C, Massow U, Vaux T, Taieb V, Deodhar A. Improved Pain, Morning Stiffness, and Fatigue With Bimekizumab in Axial Spondyloarthritis: Results From the Phase III BE MOBILE Studies. J Rheumatol. 2025 Jan 1;52(1):23-32. doi: 10.3899/jrheum.2024-0223. PMID 39406403
- [Derived] Baraliakos X, Deodhar A, van der Heijde D, Magrey M, Maksymowych WP, Tomita T, Xu H, Massow U, Fleurinck C, Ellis AM, Vaux T, Shepherd-Smith J, Marten A, Gensler LS. Bimekizumab treatment in patients with active axial spondyloarthritis: 52-week efficacy and safety from the randomised parallel phase 3 BE MOBILE 1 and BE MOBILE 2 studies. Ann Rheum Dis. 2024 Jan 11;83(2):199-213. doi: 10.1136/ard-2023-224803. PMID 37793792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in April 2019 and concluded in April 2023. Among the total of 274 participants, 254 participants were enrolled under the global study protocol by June 2021, including 16 enrolled in China. The enrolment was extended in China to achieve the target of 36 participants as agreed with the local agency and additional 20 Chinese participants were enrolled by February 2022 in the China Extension population.
Pre-assignment Details: Out of 36 Chinese participants, 16 participants were included in the analysis of global population and the results of the remaining 20 Chinese participants are reported separately as the China Extension Population. Participant Flow refers to the Randomized Set and AS0010 China Extension Participants.
Groups:
- Placebo (up to Week 16) (Global Population): Participants received placebo matched to bimekizumab 160 milligrams (mg) every 4 weeks (Q4W) subcutaneously until Week 16.
- Bimekizumab 160 mg Q4W (up to Week 16) (Global Population): Participants received bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population): At the end of the 16-week Double-Blind Treatment Period, study participants receiving placebo were re-allocated to bimekizumab treatment at Week 16. Participants from both placebo and bimekizumab arm received bimekizumab 160 mg Q4W subcutaneously from Week 16 until Week 48 during maintenance period. Participants entering the extension study received bimekizumab 160 mg Q4W subcutaneously until Week 52.
- Placebo (up to Week 16) (China Extension Population): Participants in the China Extension Population received placebo matched to bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population): Participants in the China Extension Population received bimekizumab 160 mg Q4W subcutaneously until Week 16.
- BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population): At the end of the 16-week Double-Blind Treatment Period, study participants in China Extension Population receiving placebo were re-allocated to bimekizumab treatment at Week 16. Participants from both placebo and bimekizumab arm received bimekizumab 160 mg Q4W subcutaneously from Week 16 until Week 48 during maintenance period. Participants entering the extension study received bimekizumab 160 mg Q4W subcutaneously until Week 52.
Period: Double-Blind Treatment Period:Week 1-16
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population)
Started | 126 | 128 | 0 | 11 | 9 | 0
Started Chinese Participants | 7 | 9 | 0 | 11 | 9 | 0
Completed | 118 | 126 | 0 | 11 | 9 | 0
Not Completed | 8 | 2 | 0 | 0 | 0 | 0
Not completed — Patient Compliance | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal By Study Participant | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period: Week 16-52
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population)
Started | 0 | 0 | 242 (Placebo=116+ BKZ=126 2 participants Completed the 16-Week Double-Blind Period but did not enter the Maintenance Period because of the below reason: Adverse event:) | 0 | 0 | 20
Completed | 0 | 0 | 220 | 0 | 0 | 17
Not Completed | 0 | 0 | 22 | 0 | 0 | 3
Not completed — Withdrawal By Study Participant | 0 | 0 | 12 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — COVID-19 pandemic situation & site restrictions | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non- Compliance | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set which consisted of all randomized study participants. AS0010 China Extension Participants refer to an additional randomized set recruited in China after the closure of the global study recruitment.
Groups:
- Placebo (up to Week 16) (Global Population): Participants received placebo matched to bimekizumab 160 mg Q4W subcutaneously until Week 16.
- Total: Total of all reporting groups
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | Total
Number analyzed (Participants) | 126 | 128 | 11 | 9 | 274
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 | 123 | 125 | 11 | 9 | 268
  65 - <85 | 3 | 3 | 0 | 0 | 6
  >= 85 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 55 | 7 | 2 | 125
  Male | 65 | 73 | 4 | 7 | 149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 15 | 11 | 9 | 48
  Black | 1 | 2 | 0 | 0 | 3
  White | 110 | 109 | 0 | 0 | 219
  Other/Mixed | 1 | 1 | 0 | 0 | 2
  Missing | 1 | 1 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 0 | 5
  Not Hispanic or Latino | 122 | 125 | 11 | 9 | 267
  Missing | 1 | 1 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response at Week 16
Description: ASAS40 response is defined as relative improvements of at least 40% and absolute improvement of at least 2 units in at least 3 of the 4 following components:1) Patient's Global Assessment of Disease Activity (PGADA) assessed on a scale ranging from 0 [not active] to 10 [very active], higher score=higher disease activity, 2) Spinal Pain assessed on a scale ranging from 0 [no pain] to 10 [most severe pain], higher score= higher pain intensity, 3) Bath Ankylosing Spondylitis Functional Index (BASFI) assessing participant's level of ability on a scale ranging from 0 [easy] to 10 [impossible] on 10 physical activities,4) morning stiffness, assessed as the mean of Q5 (intensity) and Q6 (duration) from the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), each assessed on a scale ranging from 0 [none / 0 hour] to 10 [very severe / 2 or more hours], higher score=higher severity; and no worsening at all in the remaining component.
Time Frame: Week 16
Population: The Randomized set consisted of all randomized study participants. AS0010 China Extension Participants refer to an additional randomized set recruited in China after the closure of the global study recruitment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
percentage of participants | 21.4 | 47.7 | 27.3 | 33.3
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.51, 95% CI 2-sided [2.00 to 6.16]

2. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 40% Response Criteria (ASAS40) Response in TNFα Inhibitor-naïve Subjects at Week 16
Description: as for outcome 1
Time Frame: Week 16
Population: The Randomized Set consisted of all randomized study participants. AS0010 China Extension Participants refer to an additional randomized set recruited in China after the closure of the global study recruitment. Participants analyzed are those from the RS who are TNFα inhibitor-naïve.
Measure: Number; unit: percentage of Participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 109 | 118 | 11 | 8
percentage of Participants | 22.9 | 46.6 | 27.3 | 37.5
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.08, 95% CI 2-sided [1.71 to 5.54]

3. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total Score at Week 16
Description: BASDAI is a well-established patient-reported endpoint assessing severity of AS symptoms. It is made of 6 items assessing severity of fatigue, spinal pain, peripheral joint pain & swelling, enthesitis, & morning stiffness (both severity and duration). Each question is rated using a numerical rating scale ranging from 0 (none) to 10 (very severe), higher score=higher symptom severity.BASDAI score is calculated by computing mean of questions 5 and 6 & adding it to sum of questions 1 to 4.This score is then divided by 5.Total BASDAI score ranges from 0=no disease activity to 10=maximal disease activity, higher score indicates higher symptom severity. A negative change reflects improvement.
Time Frame: Baseline, Week 16
Population: The Randomized Set consisted of all randomized study participants. AS0010 China Extension Participants refer to an additional randomized set recruited in China after the closure of the global study recruitment. Here, 'Number of Participants Analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 10 | 9
score on a scale | -1.55 (0.22) | -3.07 (0.21) | -2.09 (0.564) | -2.99 (0.571)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -1.51, 95% CI [-2.04 to -0.98]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.220, ANCOVA; LS Mean difference = -0.91, 95% CI 2-sided [-2.42 to 0.61]

4. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society 20% Response Criteria (ASAS20) Response at Week 16
Description: ASAS20 response is defined as relative improvements of at least 20% and absolute improvement of at least 1 unit in at least 3 of the 4 following components:1) PGADA assessed on a scale ranging from 0 [not active] to 10 [very active], higher score=higher disease activity, 2) Spinal Pain assessed on a scale ranging from 0 [no pain] to 10 [most severe pain], higher score= higher pain intensity, 3) BASFI assessing participant's level of ability on a scale ranging from 0 [easy] to 10 [impossible] on 10 physical activities, 4) morning stiffness, assessed as the mean of Q5 (intensity) and Q6 (duration) from the BASDAI, each assessed on a scale ranging from 0 [none / 0 hour] to 10 [very severe / 2 or more hours], higher score=higher severity; and no worsening at all in the remaining component.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
percentage of participants | 38.1 | 68.8 | 54.5 | 44.4
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.69, 95% CI 2-sided [2.17 to 6.26]

5. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) Partial Remission (PR) at Week 16
Description: The Assessment of SpondyloArthritis International Society partial remission (ASAS-PR) is defined as a score of less than or equal to (<=) 2 units in each of the 4 following components:1) PGADA assessed on a scale ranging from 0 [not active] to 10 [very active], higher score=higher disease activity,2) Spinal Pain assessed on a scale ranging from 0 [no pain] to 10 [most severe pain], higher score= higher pain intensity, 3) BASFI assessing participant's level of ability on a scale ranging from 0 [easy] to 10 [impossible] on 10 physical activities, and 4) morning stiffness, assessed as the mean of Q5 (intensity) and Q6 (duration) from the BASDAI scale, each assessed on a scale ranging from 0 [none / 0 hour] to 10 [very severe / 2 or more hours], higher score=higher severity.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
percentage of participants | 7.1 | 25.8 | 9.1 | 33.3
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 4.52, 95% CI 2-sided [2.06 to 9.93]

6. Secondary Outcome: Percentage of Participants With Ankylosing Spondylitis Disease Activity Score Major Improvement (ASDAS-MI) at Week 16
Description: ASDAS-MI is achieved when there is a reduction (improvement) greater or equal to (>=) 2.0 in ASDAS relative to Baseline. ASDAS is calculated by adding the 5 following components: 1) 0.121 × Neck, back or hip pain (BASDAI Q2), 2) 0.058 × Duration of morning stiffness (BASDAI Q6), 3) 0.110 × Patient's Global Assessment of Disease Activity (PGADA), 4) 0.073 × Peripheral pain/swelling in joints (BASDAI Q3), 5) 0.579 × (natural logarithm of the C-reactive protein (CRP) [mg/L] + 1). Q2, Q3 and Q6 from BASDAI and PGADA, are all assessed on a numerical scale from 0 [none / not active] to 10 [very severe / very active]. There is a minimum score of 0.980 for ASDAS (as a fixed value of 2 is assumed for values of hs-CRP below the lower limit of quantification (LLOQ)), but no defined upper score. Higher ASDAS scores reflect higher disease activity and participants achieving ASDAS-MI are considered to have a major improvement in their disease.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
percentage of participants | 7.1 | 27.3 | 9.1 | 11.1
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 5.43, 95% CI 2-sided [2.41 to 12.23]

7. Secondary Outcome: Percentage of Participants With Assessment of SpondyloArthritis International Society (ASAS) 5/6 Response at Week 16
Description: ASAS 5/6 response is defined as achieving at least 20% improvement in 5 of the following 6 components:1) PGADA assessed on a scale ranging from 0 [not active] to 10 [very active], higher score=higher disease activity, 2) Spinal Pain assessed on a scale ranging from 0 [no pain] to 10 [most intense pain], higher score=higher pain intensity,3) BASFI assessing participant's level of ability on a scale ranging from 0 [easy] to 10 [impossible] on 10 physical activities,4) morning stiffness, assessed as the mean of Q5 (intensity) and Q6 (duration) from the BASDAI scale, each assessed on a scale ranging from 0 [none/ 0 hour] to 10 [very severe / 2 or more hours], higher score=higher severity;5) spinal mobility (ie, lateral spinal flexion component of Bath Ankylosing Spondylitis Disease Metrology Index) on a scale ranging from 0 [no limitation of movement] to 10 [very severe limitation of movement] and 6) high sensitivity C-reactive protein (hs-CRP).
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
percentage of participants | 20.6 | 45.3 | 18.2 | 44.4
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.87 to 5.84]

8. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) at Week 16
Description: The BASFI is a well-established PRO measure of physical functioning used in AxSpA trials. It assesses participants' level of ability during the past week in conducting 10 physical activities on a scale ranging from 0 [easy] to 10 [impossible]. The BASFI score is the mean of the 10 item scores and ranges from 0 to 10, with lower scores indicating better physical function. A negative change in BASFI indicates improvement. The higher the negative value the better the improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 10 | 9
score on a scale | -0.91 (0.22) | -2.39 (0.21) | -0.79 (0.340) | -2.03 (0.368)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -1.48, 95% CI [-1.99 to -0.97]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.019, ANCOVA; LS Mean difference = -1.25, 95% CI 2-sided [-2.26 to -0.24]

9. Secondary Outcome: Change From Baseline in Nocturnal Spinal Pain Score Using Numeric Rating Scale (NRS) at Week 16
Description: Nocturnal spinal pain experienced by participants with axial spondyloarthritis (axSpA) was assessed on a numerical rating scale ranging from 0 (no pain) to 10 (most severe pain). A lower score indicates less pain and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 10 | 9
score on a scale | -1.71 (0.27) | -3.51 (0.25) | -2.41 (0.638) | -3.51 (0.658)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -1.80, 95% CI [-2.42 to -1.18]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.199, ANCOVA; LS Mean difference = -1.09, 95% CI 2-sided [-2.83 to 0.65]

10. Secondary Outcome: Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Total Score at Week 16
Description: The Ankylosing Spondylitis Quality of Life (ASQoL) is an 18-item PRO measure developed specifically for measuring health-related quality of life (HRQoL) in participants with ankylosing spondylitis and validated in the full spectrum of axial spondyloarthritis (axSpA). Each item is given a score of 1 for positive responses indicating impaired quality of life, and a score of 0 for negative responses. All item scores are summed to generate the total score ranging from 0 to 18 with a higher score indicating worse HRQoL. A negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 10 | 9
score on a scale | -2.30 (0.43) | -4.94 (0.42) | 0.18 (0.970) | -1.66 (0.967)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -2.63, 95% CI [-3.66 to -1.61]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.170, ANCOVA; LS Mean difference = -1.84, 95% CI 2-sided [-4.56 to 0.89]

11. Secondary Outcome: Change From Baseline in the Short Form 36-Item Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 16
Description: SF-36 is a 36-item HRQoL instrument with recall period of 4 weeks. Items are grouped into 8 domains: Physical Functioning (10 items), Role Physical (4 items), Bodily Pain (2 items), General Health (5 items), Vitality (4 items), Social Functioning (2 items), Role Emotional (3 items), Mental Health (5 items) and 1 item for Health Transition during last year. PCS and Mental Component Summary (MCS) scores are calculated from 8 domains (excluding Health Transition item). Each of SF-36 derived raw scores range from 0 to 100; higher score = better function. PCS score is calculated from 8 domain scores. It is standardized score ranging from 7.3 to 70.1, with a mean of 50 and SD of 10 in general US population, higher values = better function, and positive change reflects improvement. A PCS score mean below 47 indicates impaired physical functioning. Individual respondent's score that falls outside T-score range of 45 to 55 are outside average general US population range.
Time Frame: Baseline, Week 16
Population: Randomized Set consisted of all randomized study participants. AS0010 China Extension Participants refer to an additional randomized set recruited in China after the closure of the global study recruitment. 'Number of Participants Analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 10 | 9
T-score | 5.36 (0.79) | 9.32 (0.76) | -3.52 (2.462) | 3.75 (2.364)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = 3.96, 95% CI 2-sided [2.08 to 5.83]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.035, ANCOVA; LS Mean difference = 7.27, 95% CI 2-sided [0.60 to 13.95]

12. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Metrology Index (BASMI) at Week 16
Description: The BASMI characterizes the spinal mobility of participants with axial Spondyloarthritis (SpA) and Ankylosing Spondylitis. It is a disease-specific measure consisting of 5 clinical measures to reflect participant axial status: cervical rotation; tragus to wall distance; lateral lumbar flexion; lumbar flexion (modified Schober test); intermalleolar distance. According to the linear definition of the BASMI a score of 0 to 10 was calculated for each item based on the measurement. The mean of the 5 scores provides the total BASMI score (ranging from 0 to 10). The higher the BASMI score, the more severe the participant's limitation of movement due to their axial SpA. A negative value in BASMI change from Baseline indicates an improvement from Baseline. The higher the negative value, the better the improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 126 | 128 | 11 | 9
score on a scale | -0.11 (0.08) | -0.44 (0.08) | 0.12 (0.211) | -0.38 (0.232)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -0.33, 95% CI 2-sided [-0.52 to -0.14]
Statistical Analysis 2: Comparison: Placebo (up to Week 16) (China Extension Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population); Test type: Superiority; p = 0.086, ANCOVA; LS Mean difference = -0.50, 95% CI 2-sided [-1.07 to 0.07]

13. Secondary Outcome: Change From Baseline in the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index in the Subgroup of Participants With Enthesitis at Baseline at Week 16
Description: The Maastricht Ankylosing Spondylitis Enthesitis is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process), each scored as 0 or 1 and then summed for a possible score of 0 to 13. A higher score reflects higher severity and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: Subgroup of study participants in Randomized Set with enthesitis at Baseline (MASES index score > 0). Subgroup of study participants in China Extension Population (randomized set) with enthesitis at Baseline (MASES index score > 0).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 92 | 94 | 5 | 3
score on a scale | -1.11 (0.38) | -2.16 (0.37) | -1.35 (0.692) | -1.80 (0.871)
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p = 0.013, ANCOVA; LS Mean difference = -1.06, 95% CI 2-sided [-1.88 to -0.23]

14. Secondary Outcome: Percentage of Participants With Enthesitis-free State at Week 16 Based on the Maastricht Ankylosing Spondylitis Enthesitis (MASES) Index in the Subgroup of Participants With Enthesitis at Baseline
Description: The Maastricht Ankylosing Spondylitis Enthesitis is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process), each scored as 0 or 1 and then summed for a possible score of 0 to 13. Enthesitis free state is defined as having a MASES score of 0. A higher score reflects higher severity and a negative change represents an improvement.
Time Frame: Baseline, Week 16
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population)
Number analyzed (Participants) | 92 | 94 | 5 | 3
percentage of participants | 23.9 | 51.1 | 60.0 | 66.7
Statistical Analysis 1: Comparison: Placebo (up to Week 16) (Global Population) vs Bimekizumab 160 mg Q4W (up to Week 16) (Global Population); Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.49, 95% CI 2-sided [1.84 to 6.62]

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week Safety follow up (SFU)). TEAEs were analyzed and have been reported separately for Double-Blind Treatment Period (Safety set),Maintenance Period (MP) (Maintenance Set) and Overall Period (Safety set) which includes all participants who received BKZ 160 mg Q4W during the study. The overall period arm reports repeated TEAEs from the double blind treatment period arm and maintenance period arm. As pre-specified in SAP, Maintenance Period (MP) included AEs of Safety follow up period for participants who did not enter the open label extension or discontinued early in MP.
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68) (Week 48 last IMP intake + 20 weeks SFU)
Population: Safety Set consisted of all randomized study participants who received at least 1 dose of IMP. Maintenance Set (MS) included all study participants who have received at least 1 dose of BKZ treatment in the MP. AS0010 China Extension Participants Safety Set included all randomized study participants who received at least 1 dose of IMP. AS0010 China Extension Participants Maintenance Set included all study participants who have received at least 1 dose of BKZ treatment in the MP.
Measure: Number; unit: percentage of participants
Groups:
- Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population): Participants who received bimekizumab 160 mg Q4W subcutaneously from Day 1 up to Week 48 and participants who switched from placebo arm at Week 16 to receive bimekizumab 160 mg Q4W subcutaneously up to Week 48 were included in this group.
- Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population): Participants in the China Extension Population who received bimekizumab 160 mg Q4W subcutaneously from Day 1 up to Week 48 and participants who switched from placebo arm at Week 16 to receive bimekizumab 160 mg Q4W subcutaneously up to Week 48 were included in this group.
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population)
Number analyzed (Participants) | 126 | 128 | 242 | 244 | 11 | 9 | 20 | 20
percentage of participants | 56.3 | 62.5 | 67.8 | 75.0 | 72.7 | 100 | 80.0 | 90.0

16. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: A serious adverse event (SAE) is any untoward medical occurrence that at any dose resulted in 1) Death, 2) Life-threatening (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.), 3) Significant or persistent disability/incapacity, 4) Congenital anomaly/birth defect (including that occurring in a fetus), 5) Important medical event that, based upon appropriate medical judgment, may jeopardize the participant or participant may require medical or surgical intervention to prevent any of the above, 6) Initial inpatient hospitalization or prolongation of hospitalization. The overall period arm reports repeated SAEs from the double blind treatment period arm and maintenance period arm. As pre-specified in SAP, MP included SAEs of Safety follow up period for participants who did not enter the open label extension or discontinued early in MP.
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 68)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population)
Number analyzed (Participants) | 126 | 128 | 242 | 244 | 11 | 9 | 20 | 20
percentage of participants | 0.8 | 0 | 3.7 | 3.7 | 0 | 0 | 15.0 | 15.0

17. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Investigational Medicinal Product (IMP) During the Study
Description: TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering the 20-week SFU period). The overall period arm reports repeated events from the double blind treatment period arm and maintenance period arm. As pre-specified in SAP, MP included events of Safety follow up period for participants who did not enter the open label extension or discontinued early in MP.
Time Frame: From Baseline (Day 1) until Safety-Follow-Up (up to Week 68)
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population)
Number analyzed (Participants) | 126 | 128 | 242 | 244 | 11 | 9 | 20 | 20
percentage of participants | 4.0 | 1.6 | 2.5 | 3.3 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) until Safety Follow-Up (up to Week 68)
Description: As pre-specified in SAP, Maintenance Period (MP) included AEs of SFU period for participants who did not enter OLE or discontinued early in MP. Study participants who rolled over to OLE study did not have a SFU visit. TEAEs have been reported for Safety set (SS), MS, AS0010 China Extension Participants SS and AS0010 China Extension Participants MS. Overall Period included all participants who received BKZ 160 mg Q4W during study. Overall Period arm reports repeated TEAEs from DBTP and MP.
Arm/Group | Placebo (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) | Placebo (up to Week 16) (China Extension Population) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population)
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/128 | 0/242 | 0/244 | 0/11 | 0/9 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/126 | 0/128 | 9/242 | 9/244 | 0/11 | 0/9 | 3/20 | 3/20
Other Adverse Events (participants affected / at risk) | 30/126 | 40/128 | 94/242 | 114/244 | 8/11 | 9/9 | 13/20 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (up to Week 16) (Global Population) (N=126) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) (N=128) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) (N=242) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) (N=244) | Placebo (up to Week 16) (China Extension Population) (N=11) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) (N=9) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) (N=20) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population) (N=20)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal crusting (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abortion induced (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (up to Week 16) (Global Population) (N=126) | Bimekizumab 160 mg Q4W (up to Week 16) (Global Population) (N=128) | Bimekizumab 160 mg Q4W (Week 16 up to Week 52) (Global Population) (N=242) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (Global Population) (N=244) | Placebo (up to Week 16) (China Extension Population) (N=11) | Bimekizumab 160 mg Q4W (up to Week 16) (China Extension Population) (N=9) | BKZ 160 mg Q4W (Week 16 up to Week 52) (China Extension Population) (N=20) | Overall Period (up to Week 48 + 20 Weeks SFU): Bimekizumab 160 mg Q4W (China Population) (N=20)
Nasopharyngitis (Infections and infestations) | 6 (6) | 13 (13) | 18 (21) | 30 (34) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 9 (9) | 15 (17) | 23 (26) | 3 (5) | 1 (1) | 3 (3) | 4 (4)
Corona virus infection (Infections and infestations) | 1 (1) | 1 (1) | 17 (17) | 17 (18) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Oral candidiasis (Infections and infestations) | 0 (0) | 4 (5) | 17 (20) | 18 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (5) | 4 (6) | 10 (12) | 14 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (4) | 6 (6) | 9 (10) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 7 (8) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (3) | 2 (2) | 3 (7) | 5 (9) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3) | 4 (6) | 7 (9) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Liver function test increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (4) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligomenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (4) | 3 (5) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Axial spondyloarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT03928704/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03928704/SAP_001.pdf